CLINICAL TRIAL: NCT05947604
Title: Single Centre Open-label, Non-randomised, 3-treatment, 2-period, Pharmacokinetic Drug Interaction Study of Single Oral Dose of Acoziborole With Sequential Co-administration of Midazolam and Dextromethorphan in Healthy Male Participants
Brief Title: DDI Study of Single Oral Dose of Acoziborole With Sequential Co-administration of Midazolam and Dextromethorphan
Acronym: OXA-07
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DNDi-OXA-07-HAT
Record Dates: First submitted 2023-03-05; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Trypanosomiasis, African
MeSH Terms: conditions — Trypanosomiasis, African | interventions — Midazolam; Dextromethorphan

STUDY DESIGN:
Intervention Model Description: On Period 1, participants will receive: A single oral dose of Dextromethorphan on Day and of midazolam on Day 8.
  On Period 2, participants will receive: A single oral dose of acoziborole on Day 12, of dextromethorphan on Day 14, and of midazolam on Day 21.
  The study duration will be approximately 8 weeks:
  Screening period before the first study drug administration, Period 1 with a hospitalisation period from the day before the first dose of dextromethorphan until 24 h after the first dose of midazolam, Wash-out period: 3 days, Period 2 with a hospitalisation period from the day before the single administration of acoziborole until 24 h after the last dose of midazolam .
  End of study (EoS) visit between 7-10 days after last dose of midazolam on Period 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextromethorphan and Midazolam (Other): Drug drug interaction Dextromethorphan and Midazolam administrations
  * Dextromethorphan 15 mg syrup in fasted condition Period 1: Single oral dose of 15 mg administered on Day 1
  * Midazolam 5 mg syrup in fasted condition Period 1: Single oral dose of 5 mg administered on Day 8
  Interventions: Drug: Midazolam; Drug: Dextromethorphan
- Acoziborole, Dextromethorphan and Midazolam (Other): Drug drug interaction Acoziborole, Dextromethorphan and Midazolam administrations
  * Acoziborole 960 mg (three tablets of 320 mg) for oral route in fasted condition Period 2: single oral administration on Day 12
  * Dextromethorphan 15 mg syrup in fasted condition Period 2: Single oral dose of 15 mg administered on Day 14
  * Midazolam 5 mg syrup in fasted condition Period 2: Single oral dose of 5 mg administered on Day 21
  Interventions: Drug: Acoziborole; Drug: Midazolam; Drug: Dextromethorphan

INTERVENTIONS:
Drug: Acoziborole — Acoziborole 960 mg (three tablets of 320 mg) for oral route in fasted condition Period 2: single oral administration on Day 12
  Arms: Acoziborole, Dextromethorphan and Midazolam
Drug: Midazolam — • Midazolam 5 mg syrup in fasted condition Period 1: Single oral dose of 5 mg administered on Day 8 Period 2: Single oral dose of 5 mg administered on Day 21
Drug: Dextromethorphan — • Dextromethorphan 15 mg syrup in fasted condition Period 1: Single oral dose of 15 mg administered on Day 1 Period 2: Single oral dose of 15 mg administered on Day 14

SUMMARY:
To assess Drug drug interactions between Acoziborole and Dextromethorphan and Midazolam in healthy male volunteers.

DETAILED DESCRIPTION:
An in silico PB-PK model was developed within the simCYP software and qualified for acoziborole. This study suggested strong interactions with sensitive index substrates of CYP2D6 and CYP3A4.To validate these PB-PK model results, an open-label, non-randomised, three-treatment, one-sequence, two successive periods study with at least 3-day washout between periods was chosen to evaluate clinically the potential impact of acoziborole on plasma exposure of two different sensitive CYP substrates, DXM for CYP2D6 and midazolam for CYP3A4.

Acoziborole will be administered as a single dose, due to the long t1/2 of 360 h in healthy participants.

The SimCYP simulations showed that the best compromise to maximize the CYP2D6 inhibition and minimize the CYP3A4 induction is when DXM is given 24 to 60 h after acoziborole administration. Therefore, dextromethorphan will be given on Day 1 (in Period 1, without acoziborole) and on Day 14 in Period 2 i.e. 2 days following oral administration of acoziborole.

Based on the PB-PK simulations, the interaction between acoziborole and midazolam should be maximal around Day 8 (due to the activity CYP3A4) following acoziborole administration and sustained for several weeks after. Thus, midazolam will be given on Day 8 (in Period 1 without acoziborole) and on Day 21 in Period 2 i.e. 9 days following oral single administration of acoziborole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males.
* Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures..
* Age 18 to 55 (inclusive) years of age at the time of signing informed consent.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 as measured at screening.
* Body weight not less than 50 kg.
* Non-smokers (defined as has not used nicotine-containing products including e-cigarette for at least 3 months prior to the first dose as confirmed by cotinine test).
* Must be willing and able to communicate and participate in the whole study.
* Normal blood pressure (BP): Systolic BP (SBP) between 90 and 140 mmHg (inclusive), diastolic BP (DBP) between 45 and 90 mmHg (inclusive), measured after 10 min rest in supine position at screening and first admission (Day -1).
* A resting heart rate (HR) between 45 and 90 bpm (inclusive), measured after 10 min rest in supine position at screening and first admission (Day -1).
* ECG recording without clinically significant abnormality, including Fridericia's corrected interval between Q and T waves (QTcF) measure of ≤450 msec at screening and first admission (Day -1).
* Participants must be able to swallow multiple capsules.

Exclusion Criteria:

* Have participated in an investigational trial involving administration of any investigational compound within 90 days prior to the study dosing or 5-times the half-life of the drug tested in the previous clinical trial, whichever is longer (time calculated relative to the last dose in the previous clinical trial).
* History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption >14 units per week and (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type) as confirmed by a positive alcohol breath test at screening or any on admission to the CRW.
* Participants who do not have suitable veins for multiple venepunctures/cannulations as assessed by the Investigator or delegate at screening.
* Clinically significant abnormal clinical chemistry, haematology, urinalysis, or clinically significant abnormal physical examination findings as judged by the Investigator.
* Abnormal renal function (estimate glomerular filtration rate [eGFR] <90 mL/min).
* Confirmed positive drugs of abuse urine test result (including but not limited to, amphetamines, tetrahydrocannabinol, morphine, methamphetamine, ketamine and benzodiazepines) and at any time during the study.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
* Positive COVID test at screening and at admission of hospitalisation.
* COVID-19 full vaccination to be received less than 21 days before Day 1, or start of vaccination, or second dose or booster of vaccination planned during the study period.
* Clinically significant medical condition and/or abnormal laboratory results that could, in the opinion of the Investigator, jeopardize the participant's safety or participation in the study.
* Known serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients in the past.
* Presence or history of clinically significant allergy requiring treatment (including asthma, urticaria, clinically significant allergic rash or other severe allergic diathesis), as judged by the Investigator. Hay fever is allowed unless it is active.
* Donation or loss of greater than 400 mL of blood within the previous 3 months or more than 100 mL within 30 days before signing informed consent form (ICF) to this trial.
* Participants who are taking any prescribed drug in the 30 days before screening or require regular use of any prescription medication during the study.
* Participants who have taken, any OTC medications, including vitamins, analgesics or antacids, herbal remedies, St. John's wort or diet complements (plants and vitamins that may be used for e.g. weight control or improve digestion or for "detox"... e.g., found in the composition extracts of ginkgo biloba, aesculus, cassia, harpagophytum, curcuma, elderberry, Vitis vinifera, cypress (Cupressus sempervirens)) in the 30 days before investigational medicinal product (IMP) administration. Exceptions may apply on a case-by-case basis, if considered not to interfere with the objectives of the study, as determined by the Principal Investigator (PI).
* Use of enzyme-altering drugs (e.g. barbiturates, phenothiazines, cimetidine) within 30 days or 5 half-lives, whichever is longer, of study Day 1.
* Use of products containing quinine (e.g., tonic water), grapefruit products, pomelo products, Seville orange products, supplements containing citrus aurantium and bitter orange in the 30 days prior to study Day 1.
* CYP2D6 poor metabolizers, based on genotyping of DNA from blood samples.
* Surgery within 12 weeks prior to screening, with the exception of appendectomy or at the discretion of the Investigator for minor surgery.
* Any surgery (e.g. gastric bypass) or medical condition that may affect absorption of orally administered drugs.
* Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
To assess the effect of single dose of acoziborole on pharmacokinetics (PK) parameters (Cmax) of midazolam as a probe substrate for CYP3A4 (induction) | Up to 72 hours post drug administration
  Midazolam Cmax, plasma concentration
To assess the effect of single dose of acoziborole on pharmacokinetics (PK) parameters (Cmax) of dextromethorphan as a probe substrate for CYP2D6 (inhibition). | Up to 72 hours post drug administration
  Dextromethorphan Cmax, plasma concentration
To assess the effect of single dose of acoziborole on pharmacokinetics (PK) parameters ( AUC0-t) of midazolam as a probe substrate for CYP3A4 (induction) | Up to 72 hours post drug administration
  Midazolam AUC0-t (plasma concentration) of Period 1 and Period 2.
To assess the effect of single dose of acoziborole on pharmacokinetics (PK) parameters ( AUC0-t) of dextromethorphan as a probe substrate for CYP2D6 (inhibition). | Up to 72 hours post drug administration
  Dextromethorphan AUC0-t (plasma concentration) of Period 1 and Period 2.
To assess the effect of single dose of acoziborole on pharmacokinetics (PK) parameters (AUC0-24) of midazolam as a probe substrate for CYP3A4 (induction) | Up to 72 hours post drug administration
  Midazolam AUC0-24 (plasma concentration) of Period 1 and Period 2
To assess the effect of single dose of acoziborole on pharmacokinetics (PK) parameters (AUC0-24) of dextromethorphan as a probe substrate for CYP2D6 (inhibition). | Up to 72 hours post drug administration
  Dextromethorphan AUC0-24 of Period 1 and Period 2.

SECONDARY OUTCOMES:
To evaluate the clinical and laboratory safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to End of Study Visit, Day 31
  Frequency and cumulative incidence of treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) from time of first IMP administration (dextromethorphan on Day 1 in Period 1) to EoS visit.
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: Height | Baseline
  Vital signs for safety monitoring: Height (cm)
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: weight | Baseline and End of Study (Day 28 to Day 31)
  Vital signs for safety monitoring: Weight (Kgs)
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: Sistolic and Diastolic BP | Up to End of Study (Day 28 to Day 31)
  Vital signs for safety monitoring: Sistolic BP and Diastolic BP (mmHg)
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: respiratory rate | Up to End of Study (Day 28 to Day 31)
  Vital signs for safety monitoring: respiratory rate (breaths/minute)
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: ear body temperature | Up to End of Study (Day 28 to Day 31)
  Vital signs for safety monitoring: ear body temperature (°C).
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: 12-lead ECG Heart Rate | Up to Day 22
  12-lead electrocardiogram (ECG) Heart Rate for safety monitoring purpose. ECGs for safety purpose will be performed using the internationally recognized 12 leads with devices recorder after 10 min rest in supine position and before any blood draws. ECG will be recorded at a standard paper speed of 25 mm/s and gain of 10 mm/mV. Print-outs for each ECG will include: date, time, initials of the Investigator or its deputy.
  The ECGs will be performed in 6 × 2 leads during this study. The corresponding source data will consist of the ECG recorder paper print-outs.
  The ECGs will be read and analysed by the Investigator.
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: 12-lead ECG RR Interval | Up to Day 22
  12-lead electrocardiogram (ECG) RR Interval for safety monitoring purpose. ECGs for safety purpose will be performed using the internationally recognized 12 leads with devices recorder after 10 min rest in supine position and before any blood draws. ECG will be recorded at a standard paper speed of 25 mm/s and gain of 10 mm/mV. Print-outs for each ECG will include: date, time, initials of the Investigator or its deputy.
  The ECGs will be performed in 6 × 2 leads during this study. The corresponding source data will consist of the ECG recorder paper print-outs.
  The ECGs will be read and analysed by the Investigator.
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: 12-lead ECG QRS duration | Up to Day 22
  12-lead electrocardiogram (ECG) QRS duration for safety monitoring purpose. ECGs for safety purpose will be performed using the internationally recognized 12 leads with devices recorder after 10 min rest in supine position and before any blood draws. ECG will be recorded at a standard paper speed of 25 mm/s and gain of 10 mm/mV. Print-outs for each ECG will include: date, time, initials of the Investigator or its deputy.
  The ECGs will be performed in 6 × 2 leads during this study. The corresponding source data will consist of the ECG recorder paper print-outs.
  The ECGs will be read and analysed by the Investigator.
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: 12-lead ECG QT-interval | Up to Day 22
  12-lead electrocardiogram (ECG) QT-interval for safety monitoring purpose. ECGs for safety purpose will be performed using the internationally recognized 12 leads with devices recorder after 10 min rest in supine position and before any blood draws. ECG will be recorded at a standard paper speed of 25 mm/s and gain of 10 mm/mV. Print-outs for each ECG will include: date, time, initials of the Investigator or its deputy.
  The ECGs will be performed in 6 × 2 leads during this study. The corresponding source data will consist of the ECG recorder paper print-outs.
  The ECGs will be read and analysed by the Investigator.
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: 12-lead ECG QTcF-interval | Up to Day 22
  12-lead electrocardiogram (ECG) QTcF-interval for safety monitoring purpose. ECGs for safety purpose will be performed using the internationally recognized 12 leads with devices recorder after 10 min rest in supine position and before any blood draws. ECG will be recorded at a standard paper speed of 25 mm/s and gain of 10 mm/mV. Print-outs for each ECG will include: date, time, initials of the Investigator or its deputy.
  The ECGs will be performed in 6 × 2 leads during this study. The corresponding source data will consist of the ECG recorder paper print-outs.
  The ECGs will be read and analysed by the Investigator.
To evaluate the clinical safety of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone: 12-lead ECG PR Interval | Up to Day 22
  12-lead electrocardiogram (ECG) PR Interval for safety monitoring purpose. ECGs for safety purpose will be performed using the internationally recognized 12 leads with devices recorder after 10 min rest in supine position and before any blood draws. ECG will be recorded at a standard paper speed of 25 mm/s and gain of 10 mm/mV. Print-outs for each ECG will include: date, time, initials of the Investigator or its deputy.
  The ECGs will be performed in 6 × 2 leads during this study. The corresponding source data will consist of the ECG recorder paper print-outs.
  The ECGs will be read and analysed by the Investigator.
To evaluate the laboratory safety, Hemoglobin, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, hemoglobin, from baseline to EoS visit.
To evaluate the laboratory safety, Red blood cell count, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, Red blood cell count, from baseline to EoS visit.
To evaluate the laboratory safety, hematocrit, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, hematocrit, from baseline to EoS visit.
To evaluate the laboratory safety, white blood cells count, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, white blood cells count, from baseline to EoS visit.
To evaluate the laboratory safety, mean corpuscular volume, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, mean corpuscular volume, from baseline to EoS visit.
To evaluate the laboratory safety, mean corpuscular hemoglobin, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, mean corpuscular hemoglobin, from baseline to EoS visit.
To evaluate the laboratory safety, red cell distribution width, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, red cell distribution width, from baseline to EoS visit.
To evaluate the laboratory safety, neutrophils, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, neutrophils, from baseline to EoS visit.
To evaluate the laboratory safety, lymphocytes, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, lymphocytes, from baseline to EoS visit.
To evaluate the laboratory safety, monocytes, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, monocytes, from baseline to EoS visit.
To evaluate the laboratory safety, eosinophils, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, eosinophils, from baseline to EoS visit.
To evaluate the laboratory safety, basophils, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, basophils, from baseline to EoS visit.
To evaluate the laboratory safety, platelet count, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, platelet count, from baseline to EoS visit.
To evaluate the laboratory safety, ALP, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, ALP, from baseline to EoS visit.
To evaluate the laboratory safety, ALT, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, ALT, from baseline to EoS visit.
To evaluate the laboratory safety, AST, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, AST, from baseline to EoS visit.
To evaluate the laboratory safety, GGT, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, GGT, from baseline to EoS visit.
To evaluate the laboratory safety, CPK, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, CPK, from baseline to EoS visit.
To evaluate the laboratory safety, total bilirubin, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, total bilirubin, from baseline to EoS visit.
To evaluate the laboratory safety, direct bilirubin, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, direct bilirubin, from baseline to EoS visit.
To evaluate the laboratory safety, indirect bilirubin, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, indirect bilirubin, from baseline to EoS visit.
To evaluate the laboratory safety, total protein, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, total protein, from baseline to EoS visit.
To evaluate the laboratory safety, albumin, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, albumin, from baseline to EoS visit.
To evaluate the laboratory safety, creatinine, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, creatinine, from baseline to EoS visit.
To evaluate the laboratory safety, eGFR, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, eGFR, from baseline to EoS visit.
To evaluate the laboratory safety, fasting glucose, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, fasting glucose, from baseline to EoS visit.
To evaluate the laboratory safety, urea, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, urea, from baseline to EoS visit.
To evaluate the laboratory safety, calcium, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, calcium, from baseline to EoS visit.
To evaluate the laboratory safety, Na+, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, Na+, from baseline to EoS visit.
To evaluate the laboratory safety, K+, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, K+, from baseline to EoS visit.
To evaluate the laboratory safety, Cl-, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, Cl-, from baseline to EoS visit.
To evaluate the laboratory safety, bicarbonates, of acoziborole co-administered with midazolam and dextromethorphan as compared to administration of midazolam and dextromethorphan alone. | Up to Day 22
  Laboratory safety assessments, bicarbonates, from baseline to EoS visit.
To evaluate the Tmax of midazolam when co-administered with acoziborole. | Up to Day 22
  Time to maximum observed plasma concentration (tmax) for midazolam
To evaluate the Tmax of dextromethorphan when co-administered with acoziborole. | Up to Day 22
  Time to maximum observed plasma concentration (tmax) for dextromethorphan.
To evaluate the apparent terminal elimination half-life of midazolam when co-administered with acoziborole. | Up to Day 22
  Apparent terminal elimination half-life (t½) for midazolam
To evaluate the apparent terminal elimination half-life of dextromethorphan, when co-administered with acoziborole. | Up to Day 22
  Apparent terminal elimination half-life (t½) for dextromethorphan.
To evaluate the AUC0-∞ of midazolam when co-administered with acoziborole. | Up to Day 22
  AUC0-∞ for midazolam
To evaluate the AUC0-∞ of dextromethorphan when co-administered with acoziborole. | Up to Day 22
  AUC0-∞ for dextromethorphan.
To evaluate the Acoziborole plasma concentrations when co-administered with midazolam and dextromethorpharm | Up to Day 22
  Acoziborole plasma concentrations
To evaluate the Cmax of midazolam's metabolite, 1'hydroxy-midazolam, when co-administered with acoziborole. | Up to Day 22
  1'-hydroxy-midazolam: Cmax for Period 1 and Period 2.
To evaluate the Tmax of midazolam's metabolite, 1'hydroxy-midazolam, when co-administered with acoziborole. | Up to Day 22
  1'-hydroxy-midazolam: tmax for Period 1 and Period 2.
To evaluate the AUC0-24 of midazolam's metabolite, 1'hydroxy-midazolam, when co-administered with acoziborole. | Up to Day 22
  1'-hydroxy-midazolam:AUC0-24 for Period 1 and Period 2.
To evaluate the AUC0-t of midazolam's metabolite, 1'hydroxy-midazolam, when co-administered with acoziborole. | Up to Day 22
  1'-hydroxy-midazolam: AUC0-t for Period 1 and Period 2.
To evaluate the t½ of midazolam's metabolite, 1'hydroxy-midazolam, when co-administered with acoziborole. | Up to Day 22
  1'-hydroxy-midazolam: t½ for Period 1 and Period 2.
To evaluate the AUC0-∞ of midazolam's metabolite, 1'hydroxy-midazolam, when co-administered with acoziborole. | Up to Day 22
  1'-hydroxy-midazolam: AUC0-∞ for Period 1 and Period 2.
To evaluate the Cmax of dextromethorphan's metabolite, dextrorphan (DXO), when co-administered with acoziborole. | Up to Day 22
  DXO: Cmax for Period 1 and Period 2.
To evaluate the Tmax of dextromethorphan's metabolite, dextrorphan (DXO), when co-administered with acoziborole. | Up to Day 22
  DXO: tmax for Period 1 and Period 2.
To evaluate the AUC0-24 of dextromethorphan's metabolite, dextrorphan (DXO), when co-administered with acoziborole. | Up to Day 22
  DXO: AUC0-24 for Period 1 and Period 2.
To evaluate the AUC0-t of dextromethorphan's metabolite, dextrorphan (DXO), when co-administered with acoziborole. | Up to Day 22
  DXO: AUC0-t for Period 1 and Period 2.
To evaluate the t½ of dextromethorphan's metabolite, dextrorphan (DXO), when co-administered with acoziborole. | Up to Day 22
  DXO: t½ for Period 1 and Period 2.
To evaluate the AUC0-∞ of dextromethorphan's metabolite, dextrorphan (DXO), when co-administered with acoziborole. | Up to Day 22
  DXO: AUC0-∞ for Period 1 and Period 2.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Ng Shi Min, Principal Investigator — Clinical Research Center (CRC) Ampang Hospital
Locations (1):
- Clinical Research Center (CRC) Ampang Hospital, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT05947604/Prot_000.pdf